CLINICAL TRIAL: NCT01146535
Title: Pilot Study of Interferon Alpha Lozenges Plus Oseltamivir in the Treatment of Influenza A Infection
Brief Title: Interferon Alpha Lozenges Plus Oseltamivir for Influenza Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Collaborators: CytoPharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QCR09025
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Influenza A Virus Infection
Keywords: interferon-alpha; oseltamivir; drug therapy, combination; influenza; therapies, investigational
MeSH Terms: conditions — Influenza, Human | interventions — Interferon-alpha; Oseltamivir; Maltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interferon-alpha (Experimental): Interferon-alpha
  150 IU lozenges bid for 5 days
  Interventions: Drug: Interferon-alpha; Drug: Oseltamivir
- maltose (Placebo Comparator): maltose
  200 mg maltose lozenges bid for 5 days
  Interventions: Drug: Oseltamivir; Other: maltose

INTERVENTIONS:
Drug: Interferon-alpha — 150 IU lozenges bid for 5 days
  Other Names: IFN lozenge
  Arms: Interferon-alpha
Drug: Oseltamivir — 75 mg capsules bid for 5 days
  Other Names: Tamiflu
Other: maltose — 200 mg maltose lozenges bid for 5 days
  Other Names: placebo
  Arms: maltose

SUMMARY:
This study aims to evaluate the safety and effect of interferon-alpha lozenges when used in combination with oseltamivir (Tamiflu) to treat influenza.

ELIGIBILITY:
Inclusion Criteria:

* fever >=38C
* one or more respiratory symptoms (e.g. cough, rhinorrhea or sore throat) plus one or more constitutional symptoms (e.g. chills, headache, malaise and myalgias)of < 48 hours' duration
* body weight > 40 kg
* positive for influenza A (nasal swab rapid test)

Exclusion Criteria:

* pregnancy/lactation
* history of depression or psychiatric disorders
* history of conditions that could complicate flu infection, such as chronic pulmonary, cardiac, renal, or metabolic disorders
* use of immunosuppressive therapy
* HIV infection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Resolution of fever and flu symptoms | Days 1-5
  Time to resolution of influenza symptoms defined as all flu symptoms scored as <=1 and change in viral load (RT-PCR).

SECONDARY OUTCOMES:
Clinical response | Day 3 and Day 6
  Proportion of clinical responders on Day 3 and Day 6: defined as no fever (oral temperature < 38 °C and no subjective fever) AND resolution of influenza illness (all flu symptoms and interference scored as ≤ 1).
Proportion of poor responders | Day 3 and Day 6
  Proportion of poor responders on both Day 3 and Day 6: defined as subjects with fever (oral temperature ≥ 38 °C or any record of subjective fever) OR unresolved influenza illness (1 or more flu symptoms/interferences scored as > 1).
Time to resolution of fever | Days 1-5
  Time to bring down a fever (oral temperature < 38 °C and no subjective fever) and time to return to afebrile state (oral temperature ≤ 37.2 °C and no subjective fever).
Time to resolution of influenza illness | Days 1-5
  Time to resolution of influenza illness (all flu symptoms and interference scored as ≤ 1) as reported by the subject.
Symptom improvement | Days 1-5
  Improvement of influenza symptoms and level of interference of disease during treatment period as reported by the subject.
OTC medication usage | Days 1-5
  Proportion of use of the OTC medication for fever or influenza symptoms.
Physician visits | Days 6-10
  Rate of requirement for additional physician visits within 5 days treatment period.
Treatment failure | Days 1-28
  Rate of treatment failure including hospitalization due to disease progression prior to Day 29.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Chang Gung Medical Foundation, LinKou Branch, Guishan, Taoyuan County
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Zuoying District
  - Show-Chwan Memorial Hospital, Changhua
  - Taiwan Municipal Hospital, Tainan